CLINICAL TRIAL: NCT02300792
Title: The Effects of Honey, as a Dietary Supplement in Children With Hepatitis A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mamdouh abdulmaksoud abdulrhman, professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/013
Record Dates: First submitted 2014-11-19; First posted 2014-11-25 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Hepatitis A
Keywords: honey, hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Honey; Molasses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- honey (Active Comparator): Each patient in the honey group (group 1) took oral honey in a dose of 5 ml/kg/day (with a maximum dose of 150 ml/day) for four weeks.
  Interventions: Dietary Supplement: honey; Dietary Supplement: molasses
- molasses (Placebo Comparator): Each patient in the molasses (placebo) group (group 1) took molasses in a dose of 5 ml/kg/day (with a maximum dose of 150 ml/day) for four weeks.
  Interventions: Dietary Supplement: honey; Dietary Supplement: molasses

INTERVENTIONS:
Dietary Supplement: honey — Each patient in the intervention group (group 1) took oral honey in a dose of 5 ml/kg/day (with a maximum dose of 150 ml/day) for four weeks.
Dietary Supplement: molasses — Each patient in the molasses (placebo) group took 5 ml molasses/kg/day for four weeks, with a maximum of 150 ml/day
  Other Names: placebo

SUMMARY:
This study is a randomized, placebo controlled, double-blinded clinical trial, which included 50 children with hepatitis A. They were of both sexes and their age ranged from 2 to 18 years. The patients were randomly assigned into one of two groups; each consisted of 25 children. Each patient in the intervention group (group 1) took oral honey in a dose of 5 ml/kg/day (with a maximum dose of 150 ml/day) for four weeks, whereas patients of the placebo group (group 2) took placebo in the form of molasses. The main outcome measure was the recovery time defined as the number of days from the start of the intervention to subsidence of symptoms and signs of hepatitis and return of liver transaminases to their normal levels.

DETAILED DESCRIPTION:
This study is a randomized, placebo controlled double-blinded clinical trial, which was conducted at the Children's Hospital of Ain Shams university during the period from November 2013 to May 2014. Eligible patients were previously healthy children of both sexes, aged 2 to 18 years, who developed manifestations of acute hepatitis. Patients with diabetes mellitus (DM), chronic liver diseases, autoimmune disorders, renal disorders, neurologic diseases or malignancy were excluded from the study. Eighty nine eligible patients were recruited from the outpatient Clinic of the Children's Hospital of Ain Shams university and were subjected to history taking, physical examination and laboratory investigations in the form of serum alanine aminotransferase (ALT), serum aspartate aminotransferase (AST), serum gamma gultamyltransferase (GGT), serum bilirubin (total and direct) and assay for Hepatitis A Virus IgM (HAV IgM). Only patients who had positive HAV IgM were candidates for this study. They were seventy six patients who were randomly assigned following simple randomisation procedure (computerized random numbers) to 1 of 2 groups with a 1:1 allocation ratio.

During the study, a total of twenty six patients were excluded; nine patients stopped the trial because they refused to repeat blood sampling for investigations, six patients were not compliant to honey intake and ten patients lost follow up. Fifty patients, thus completed the study protocol and were included in the final analysis.

Assuming the mean duration of the acute illness is 6 weeks and the mean (±SD) duration of acute illness in the intervention group is 4 (±2), a total sample size of 42 patients (21 per group) is required to have a statistical power of 90% (alpha=0. 05). Post- hoc test was used for power calculation.

Each patient in the intervention group (group 1) took oral honey in a dose of 5 ml/kg/day (with a maximum dose of 150 ml/day) for four weeks. The dose of honey was empirical.

Each patient in the placebo group (group 2) took 5 ml molasses/kg/day; with a maximum of 150ml/day. Molasses is a honey-like substance made when cane sugar is processed. It contains no fat and is composed mainly of sucrose, besides some fructose and glucose.

The main outcome measure was the recovery time defined as the number of days from the start of the intervention to subsidence of symptoms and signs of hepatitis and return of liver transaminases to their normal levels. The main symptoms and signs of hepatitis A are fever, anorexia, nausea, vomiting, abdominal pain, dark urine, clay-colored stools and jaundice. Physical examination focused on general condition, vital data, jaundice, hepatosplenomegaly and ascites. The laboratory work up consisted of measurements of ALT, AST and GGT by kinetic method, measurement of total and direct bilirubin levels by colorimetric method, and assay of Anti-HAV IgM by ELISA.

Clinical and laboratory evaluation of each patient was done at baseline (0), 2nd week and 4th week (endpoint).

ELIGIBILITY:
Inclusion Criteria:

Previously healthy children who have Hepatitis A.They were of both sexes and aged 2 to 18 years.

Exclusion Criteria:

Patients with diabetes mellitus (DM), chronic liver diseases, autoimmune disorders, renal disorders, neurologic diseases or malignancy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
the recovery time defined as the number of days from the start of the intervention to subsidence of symptoms and signs of hepatitis and return of liver transaminases to their normal levels. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh A Abdulrhman, Professor, Principal Investigator — Ain Shams University